CLINICAL TRIAL: NCT07031934
Title: Investigation of the Relationships Between Core Muscle Endurance, Pelvic Oscillations and Pelvic Width in Athletes and Sedentaries
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Fırat Kara, PhD Student, Gazi University
Other Study IDs: GAZIU-FTR-FK-002
Record Dates: First submitted 2025-06-02; First posted 2025-06-22 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Core Muscle Endurance; Athlete; Sedentary
Keywords: core muscle endurance; pelvis width; pelvis oscillation; sedentary; athlete
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes Group: group of athlete individuals
- Sedentaries Group: group of sedentary individuals

SUMMARY:
The aim of this study was to investigate the relationships between pelvic oscillation, pelvic width and core muscle endurance between healthy athletes and sedentary subjects.

DETAILED DESCRIPTION:
There are many physical, physiological, psychological and sociological differences between athletes and sedentary individuals. These differences are evident due to the motoric characteristics brought about by the sports they do. While the differences revealed by the studies in the literature are in a relationship among themselves, this has an effect on the sportive performance of the person.

Core muscles are the muscles that provide both stability and mobility of the trunk in which local and global muscles work in coordination. The endurance and strength of the core muscles affect not only trunk movements but also distal extremity movements and functionality. The endurance of the core muscles, which is important for movement and balance in athletes and sedentary individuals, can also be the cause of some injuries when it is deficient.

During gait, the pelvis makes sinusoidal up-and-down movements in the frontal and sagittal planes and rotational movements in the transverse plane. These movements are provided by the local and global muscles surrounding the pelvis and hip joint. Reduction of pelvic oscillations in the normal gait pattern may lead to decreased energy expenditure and increased muscle force production. Pelvic oscillations should be sufficient and pelvic control should be appropriate for walking, running, activities of daily living and sportive performance to be correct and economical. As a result of studies showing that pelvic width has effects on the physical activities of individuals, anatomical anthropometric characteristics of the pelvis also have an effect on energy consumption in athletes and sedentary individuals.

When the literature was reviewed in this direction, no study was found that examined the relationship between core muscle endurance, pelvic swing and pelvic width in athletes and sedentary individuals. In athletes, holistic performance parameters and anthropometric characteristics or adaptations are important for the efficiency of sports. Likewise, in sedentary individuals, these characteristics are important for achieving activities of daily living. Our study is planned to examine the relationships between core muscle endurance, pelvic swing and pelvic width in athletes and sedentary individuals and to make a comparison between these two groups. As a result of the study, this gap in the literature will be filled and the relationship between core muscle endurance, pelvic swing and pelvic width of athletes will be examined and possible differences between athletes and sedentary individuals will be revealed.

ELIGIBILITY:
For Athletes Inclusion Criteria:

* Training at least 3 days a week
* Being a licensed athlete
* To be between the ages of 18-35
* Not having any locomotor system disorder
* Volunteering to participate in the study

For Sedentaries Inclusion Criteria:

* Not practicing any sport
* Not being a licensed athlete
* To be between the ages of 18-35
* Not having any locomotor system disorder
* Volunteering for the study

Exclusion Criteria:

* Chronic pain in the lumbopelvic region
* History of lumbopelvic and coronary surgery
* Having a locomotor system disorder
* Being a disabled athlete or disabled individual
* Systemic or metabolic disease

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Athletes registered to sports federations in the cities of Ankara and Kayseri
  * University students in the cities of Ankara and Kayseri
Sampling Method: Non-Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2025-06-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-12-07 (Actual)

PRIMARY OUTCOMES:
Core Muscle Endurance | four weeks
  Evaluation of core muscle endurance will be performed with the Wall Sit Hold, which have proven to be effective in the literature. In the Wall Sit Hold test, individuals will be asked to stand in a squat position with the hip and knee flexed and the back in full contact with the wall and to lift their right or left foot up and wait. The hold time will be recorded in seconds. 3 trials will be made for each foot and the results will be averaged. The higher the data obtained, the higher the core muscle endurance.
Core Muscle Endurance | four weeks
  In the Trunk Flexion Hold test, the individuals will be asked to sit on their hips and extend their upper body to the feet and knees that are lifted off the floor and wait in this position. The holding time will be recorded in seconds. The hold time will be recorded in seconds. 3 trials will be made for each foot and the results will be averaged. The higher the data obtained, the higher the core muscle endurance.
Core Muscle Endurance | four weeks
  In the Horizontal Trunk Hold test, individuals will be asked to extend both arms to the side without bending their back and wait in the crawling position. The hold time will be recorded in seconds. 3 trials will be made for each foot and the results will be averaged. The higher the data obtained, the higher the core muscle endurance.

SECONDARY OUTCOMES:
Pelvis Width | four weeks
  Pelvic width will be measured with an anthropometric measurement set caliper between the iliac cristae over both thoracentor major and both Sias of the participant lying on the bed on the back. The pelvic width will be recorded in cm without any belt or pants.
Pelvis Oscillations | four weeks
  Pelvic sway assessment will be performed with a device called GYKO, which includes a gyroscope, magnetometer and accelerometer. In this assessment, the individual will be asked to walk normally on flat ground for 10 m after the device is connected to the level of the proc. spinosus of the lumbar 3-5th vertebrae with a waist belt. The device, which is connected to the computer via Bluetooth, will generate data by recording the oscillations of the pelvis in square centimeters (cm2) throughout the walk. It will also record anterior-posterior home medial-lateral oscillations.

CONTACTS AND LOCATIONS:
Overall Officials: Fırat Kara, Phd Student, Principal Investigator — Nuh Naci Yazgan University
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No